CLINICAL TRIAL: NCT05384028
Title: Effects of Nurse-led Case Management Based on Multidisciplinary Collaboration in the Whole Course Prevention and Control of Acute Myocardial Infarction
Brief Title: Effects of Nurse-led Case Management Based on Prevention and Control of Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XJTU1AF2022LSK-169
Record Dates: First submitted 2022-04-26; First posted 2022-05-20 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; case management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients in the experimental group will receive full-course case management from a multidisciplinary team from admission to 6 months after discharge
  Interventions: Other: Nurse -led case management
- Control (Active Comparator): Patients in the control group will receive routine inpatient care and post-discharge follow-up management
  Interventions: Other: Routine inpatient care and post-discharge follow-up management

INTERVENTIONS:
Other: Nurse -led case management — This study would apply case management to the whole course management of AMI patients from admission to 6 months after discharge. Pharmacists, nutritionists, rehabilitation specialists and psychiatrists led by nurse would take the initiative to conduct individualized assessment and health guidance, and case managers would participate in the whole process of inpatient diagnosis and treatment. Coordinating multidisciplinary medical resources to jointly implement diagnosis and treatment and rehabilitation for patients can improve the quality of care.
  Arms: Experimental
Other: Routine inpatient care and post-discharge follow-up management — Patients in the control group will receive routine inpatient care and post-discharge follow-up management
  Arms: Control

SUMMARY:
Acute Myocardial Infarction (AMI) is a major disease that endangers people's health China. At present, clinical emphasis is given to "treatment" rather than "prevention", and a large number of AMI patients are hospitalized repeatedly without systematic and standardized health management after acute stage, falling into a vicious circle of "treatment without recovery". Nurse-led case management based on multidisciplinary collaboration is a new mode of disease management. In 1994, the United States took the lead in applying case management to the acute and chronic care system, providing comprehensive care services and promoting comprehensive recovery through multidisciplinary collaboration led by case managers. At present, the case management model of cardiovascular disease in Europe and the United States has been mature, but it is still in the exploratory stage in China. Through the establishment and application of nurse-led AMI case management program based on multidisciplinary collaboration, this study wants to establish a novel, standardized, and easy to popularize AMI whole-course prevention and control mode, providing theoretical and research basis for AMI disease management.

DETAILED DESCRIPTION:
There are few domestic studies on cardiovascular disease case management in China, and the studies mainly aimed at the application of case management in out-of-hospital follow-up management. At present, there has been no reports on nurse-led the multidisciplinary whole course case management of AMI patients from admission to discharge, diagnosis and treatment, rehabilitation and secondary prevention. This study would apply case management to the whole course management of AMI patients from admission to 6 months after discharge. Pharmacists, nutritionists, rehabilitation specialists and psychiatrists coordinated by nurse would take the initiative to conduct individualized assessment and health guidance, and case managers would participate in the whole process of inpatient diagnosis and treatment. Coordinating multidisciplinary medical resources to jointly implement diagnosis and treatment and rehabilitation for patients can save medical costs and improve the quality of care.

ELIGIBILITY:
Inclusion Criteria:

* In line with the diagnosis of Chinese 2019 Guidelines for AMI. Age greater than or equal to 18 years old and less than or equal to 75 years old Patients have clear consciousness and agree to participate in this study.

Exclusion Criteria:

* Verbal communication disorders. Patients have a clear history of allergic constitution, and have allergies or intolerance to the drugs recommended by the guidelines (including antiplatelet drugs, ẞ receptor blockers, statins, various antihypertensive and hypoglycemic drugs, etc.).

Patients have severe heart, brain, liver, kidney, motor dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
The 36-item Short Form Health Survey for HRQoL | from baseline to 6 months after discharge
  Health-related quality of life
Coronary artery disease self-management scale for self-management behaviors | from baseline to 6 months after discharge
  Self-management behaviors
the numbers of unplanned readmission | Through study completion, within 6 months post discharge
  Unplanned readmission
the number of deaths from cardiac causes | Through study completion,within 6 months post discharge
  Deaths from cardiac causes

SECONDARY OUTCOMES:
the numbers of no smoking | from baseline to 6 months after discharge
  Smoking
systolic and diastolic blood pressure （mmHg） | from baseline to 6 months after discharge
  Blood Pressure.
Glycated hemoglobin A1c （%） | from baseline to 6 months after discharge
  Collect fasting venous blood to measure glycosylated hemoglobin A1c
Body mass index (BMI)，kg/m2 | from baseline to 6 months after discharge
  Measure weight and height，then weight and height will be combined to report BMI in kg/m^2
Low-density lipoprotein （mmol/L） | from baseline to 6 months after discharge
  Collect fasting venous blood to measure low-density lipoprotein
Exercise time every week （min） | from baseline to 6 months after discharge
  Inquire the exercise time per week

CONTACTS AND LOCATIONS:
Locations (1):
- Jingwen Hu, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sunamura M, Ter Hoeve N, Geleijnse ML, Steenaard RV, van den Berg-Emons HJG, Boersma H, van Domburg RT. Cardiac rehabilitation in patients who underwent primary percutaneous coronary intervention for acute myocardial infarction: determinants of programme participation and completion. Neth Heart J. 2017 Nov;25(11):618-628. doi: 10.1007/s12471-017-1039-3. PMID 28917025
- [Background] Pocock S, Bueno H, Licour M, Medina J, Zhang L, Annemans L, Danchin N, Huo Y, Van de Werf F. Predictors of one-year mortality at hospital discharge after acute coronary syndromes: A new risk score from the EPICOR (long-tErm follow uP of antithrombotic management patterns In acute CORonary syndrome patients) study. Eur Heart J Acute Cardiovasc Care. 2015 Dec;4(6):509-17. doi: 10.1177/2048872614554198. Epub 2014 Oct 9. PMID 25301783
- [Background] Puymirat E, Bonaca M, Iliou MC, Tea V, Ducrocq G, Douard H, Labrunee M, Plastaras P, Chevallereau P, Taldir G, Bataille V, Ferrieres J, Schiele F, Simon T, Danchin N; FAST-MI investigators. Outcome associated with prescription of cardiac rehabilitation according to predicted risk after acute myocardial infarction: Insights from the FAST-MI registries. Arch Cardiovasc Dis. 2019 Aug-Sep;112(8-9):459-468. doi: 10.1016/j.acvd.2019.04.002. Epub 2019 May 22. PMID 31126738
- [Background] Li J, Dharmarajan K, Bai X, Masoudi FA, Spertus JA, Li X, Zheng X, Zhang H, Yan X, Dreyer RP, Krumholz HM. Thirty-Day Hospital Readmission After Acute Myocardial Infarction in China. Circ Cardiovasc Qual Outcomes. 2019 May;12(5):e005628. doi: 10.1161/CIRCOUTCOMES.119.005628. PMID 31092023
- [Background] DeBusk RF, Miller NH, Superko HR, Dennis CA, Thomas RJ, Lew HT, Berger WE 3rd, Heller RS, Rompf J, Gee D, Kraemer HC, Bandura A, Ghandour G, Clark M, Shah RV, Fisher L, Taylor CB. A case-management system for coronary risk factor modification after acute myocardial infarction. Ann Intern Med. 1994 May 1;120(9):721-9. doi: 10.7326/0003-4819-120-9-199405010-00001. PMID 8147544
- [Background] Berra K. Does nurse case management improve implementation of guidelines for cardiovascular disease risk reduction? J Cardiovasc Nurs. 2011 Mar-Apr;26(2):145-67. doi: 10.1097/JCN.0b013e3181ec1337. PMID 21076315
- [Background] Stafford RS, Berra K. Critical factors in case management: practical lessons from a cardiac case management program. Dis Manag. 2007 Aug;10(4):197-207. doi: 10.1089/dis.2007.103624. PMID 17718658
- [Background] O'Neill JL, Cunningham TL, Wiitala WL, Bartley EP. Collaborative hypertension case management by registered nurses and clinical pharmacy specialists within the Patient Aligned Care Teams (PACT) model. J Gen Intern Med. 2014 Jul;29 Suppl 2(Suppl 2):S675-81. doi: 10.1007/s11606-014-2774-4. PMID 24715403
- [Background] Huntley AL, Thomas R, Mann M, Huws D, Elwyn G, Paranjothy S, Purdy S. Is case management effective in reducing the risk of unplanned hospital admissions for older people? A systematic review and meta-analysis. Fam Pract. 2013 Jun;30(3):266-75. doi: 10.1093/fampra/cms081. Epub 2013 Jan 12. PMID 23315222
- [Background] Ensign CM, Hawkins SY. Improving Patient Self-Care and Reducing Readmissions Through an Outpatient Heart Failure Case Management Program. Prof Case Manag. 2017 Jul/Aug;22(4):190-196. doi: 10.1097/NCM.0000000000000232. No abstract available. PMID 28557879
- [Background] Tosun N, Akbayrak N. Global case management: using the case management model for the care of patients with acute myocardial infarction in a military hospital in Turkey. Lippincotts Case Manag. 2006 Jul-Aug;11(4):207-15. doi: 10.1097/00129234-200607000-00004. PMID 16926693
- [Background] Chen YC, Chang YJ, Tsou YC, Chen MC, Pai YC. Effectiveness of nurse case management compared with usual care in cancer patients at a single medical center in Taiwan: a quasi-experimental study. BMC Health Serv Res. 2013 May 31;13:202. doi: 10.1186/1472-6963-13-202. PMID 23725552